CLINICAL TRIAL: NCT05126680
Title: Vascular-Fit: Efficacy of an In-hospital Physical Exercise Program on Functional Capacity and Quality of Life in Patients With Peripheral Artery Disease
Brief Title: Moderate Intensity Functional Training as Adjuvant Treatment in Patients With Peripheral Arterial Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European University Miguel de Cervantes (Other)
Collaborators: Hospital Clínico Universitario de Valladolid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI-DOC001-PAD
Record Dates: First submitted 2021-11-08; First posted 2021-11-19 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Peripheral Arterial Disease; Intermittent Claudication
Keywords: Peripheral arterial disease; Supervised exercise therapy; Functional training; Intermittent claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent treadmill walking exercise and moderate intensity functional training (Experimental): Subjects belonging to this group perform a 12-week supervised exercise therapy consisted of intermittent treadmill walking exercise and moderate intensity functional training.
  Interventions: Other: Supervised exercise therapy: intermittent treadmill walking exercise and moderate intensity functional training
- Intermittent treadmill walking exercise (Active Comparator): Subjects belonging to this group perform a 12-week supervised exercise therapy consisted of intermittent treadmill walking exercise.
  Interventions: Other: Supervised exercise therapy: intermittent treadmill walking exercise

INTERVENTIONS:
Other: Supervised exercise therapy: intermittent treadmill walking exercise and moderate intensity functional training — Subjects will perform a 12-week supervised exercise therapy program based on intermittent treadmill walking exercise (15-30 min.) and moderate intensity functional training (MIFT) (15 min.). In intermittent treadmill walking exercise, the speed and incline of treadmill will be adjusted that patients achieve moderate claudication pain in the time interval between 3 and 5 min. In MIFT, subjects must complete in 15 min. the highest number of repetitions / rounds possible (AMRAP) to a circuit composed of 6 global functional exercises from which they performed 10 repetitions with a rating of perceived exertion (RPE) of 5-7 on a 1 to 10 scale in each exercise.
  Arms: Intermittent treadmill walking exercise and moderate intensity functional training
Other: Supervised exercise therapy: intermittent treadmill walking exercise — Subjects will perform a 12-week supervised exercise therapy program based on intermittent treadmill walking exercise (30-45 min.). In intermittent treadmill walking exercise, the speed and incline of treadmill will be adjusted that patients achieve moderate claudication pain in the time interval between 3 and 5 min.
  Arms: Intermittent treadmill walking exercise

SUMMARY:
Traditional aerobic training and muscle resistance ('strength') training have been shown to be effective for improving functional and health-related quality of life (HRQoL) outcomes in peripheral arterial disease (PAD). However, the transfer of the current resistance exercise modes proposed to other activities of daily living (ADLs) is questionable. Moderate intensity functional training (MIFT) has emerged with the aim of achieving cardiovascular and neuromuscular adaptations simultaneously with functional exercises typical of ADLs. The effect of MIFT in patients with PAD is not yet known. Our purpose is to verify the influence of the combination of intermittent treadmill walking exercise with MIFT compared with intermittent treadmill walking exercise on functional capacity, HRQoL, biochemical and hemodynamic parameters in patients with PAD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with PAD in grade IIa (Leriche-Fontaine Classification).

Exclusion Criteria:

* Subjects with dementia.
* Institutionalized Subjects in social health centers.
* Subjects with recent major surgery in the last year or lower limb amputations.
* Subjects with revascularization surgery of the lower extremities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Six-Minute Walk Test | 0 weeks, 6 weeks and 12 weeks.
  Changes in maximum walking distance (MWD) and claudication onset distance (COD).
Moderate intensity functional training Test | 0 weeks, 6 weeks and 12 weeks.
  Changes in number of rounds/repetitions and total workload.
Short Form-36 Health Survey (SF-36) | 0 weeks, 6 weeks and 12 weeks.
  Changes in the eight domains of health status.
Vascular Quality of Life Questionnaire-6 (VascuQol-6) | 0 weeks, 6 weeks and 12 weeks.
  Changes in total punctuation of questionnaire.

SECONDARY OUTCOMES:
Biochemical analysis | 0 weeks, 6 weeks and 12 weeks.
  Changes in complete lipid profile
Biochemical analysis | 0 weeks, 6 weeks and 12 weeks.
  Changes in lactate dehydrogenase
Biochemical analysis | 0 weeks, 6 weeks and 12 weeks.
  Changes in c-reactive protein
Biochemical analysis | 0 weeks, 6 weeks and 12 weeks.
  Changes in tumor necrosis factor alpha
Biochemical analysis | 0 weeks, 6 weeks and 12 weeks.
  Changes in serum apolipoproteins
Biochemical analysis | 0 weeks, 6 weeks and 12 weeks.
  Analysis of the complete oxidative profile
Hemodynamic measurements | 0 weeks, 6 weeks and 12 weeks.
  Changes in mean, systolic and diastolic blood pressure.
Hemodynamic measurements | 0 weeks, 6 weeks and 12 weeks.
  Changes in flow-mediated dilation of the brachial artery
Hemodynamic measurements | 0 weeks, 6 weeks and 12 weeks.
  Changes in ankle-brachial index
Hemodynamic measurements | 0 weeks, 6 weeks and 12 weeks.
  Changes in pulse wave velocity

CONTACTS AND LOCATIONS:
Locations (1):
- European University Miguel of Cervantes, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Penin-Grandes S, Lopez-Ortiz S, de la Fuente Gomez M, Pinto-Fraga J, Lista S, Maroto-Izquierdo S, Lucia A, Del Rio Sola ML, Martin-Hernandez J, Santos-Lozano A. Move Better, Live Better: A Novel Supervised Combined Training for Peripheral Arterial Disease: A Quasi-experimental Approach. Am J Phys Med Rehabil. 2025 Sep 1;104(9):771-779. doi: 10.1097/PHM.0000000000002706. Epub 2025 Jan 6. PMID 39792377